CLINICAL TRIAL: NCT02827734
Title: Evaluation of Novel Lung Function Parameters in Patients With Interstitial Lung Disease (ILD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Dr. Frederik Trinkmann, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: MBW-ILD
Record Dates: First submitted 2016-06-30; First posted 2016-07-11 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Healthy Controls; Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis; Non-specific Interstitial Pneumonia; Sarcoidosis; Granulomatosis With Polyangiitis (Wegener's Disease)
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis; Sarcoidosis; Granulomatosis with Polyangiitis | interventions — Plethysmography, Whole Body

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- interstitial lung disease: patients with known or suspected ILD such as idiopathic pulmonary fibrosis, non-specific interstitial pneumonia, sarcoidosis, granulomatosis with polyangiitis
  Interventions: Device: multiple breath washout tests; Device: impulse oscillometry; Device: body plethysmography
- pulmonary healthy controls: patients without known or suspected pulmonary disease
  Interventions: Device: multiple breath washout tests; Device: impulse oscillometry; Device: body plethysmography

INTERVENTIONS:
Device: multiple breath washout tests
Device: impulse oscillometry
Device: body plethysmography

SUMMARY:
Current diagnostic tools used in interstitial lung disease (ILD) do not meet the challenges set by the complex pathophysiology of this heterogenous group. The investigators therefore aimed to evaluate novel or not widely used diagnostic approaches for the detection and therapeutic monitoring of patients with various ILDs.

ELIGIBILITY:
Inclusion Criteria:

* known or suspected interstitial lung disease

Exclusion Criteria:

* pregnancy
* inability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with indication for routine lung function testing
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
lung clearance index (LCI) as determined by multiple breath washout | 30 minutes
airway resistance and reactance (R5, X5, R-D5-20) as determined by impulse oscillometry | 30 minutes

SECONDARY OUTCOMES:
repeatability of lung clearance index (LCI) | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsmedizin Mannheim, Mannheim, Deutschland, Germany

IPD SHARING:
Plan to Share IPD: No